CLINICAL TRIAL: NCT02624856
Title: Prospective, Randomized, Double-Blinded, Allocation Concealed Study Comparing the Efficacy of Liposomal Bupivacaine Over Standard Bupivacaine Plus Dexamethasone in Quadriceps Sparing Femoral Nerve Block and Wound Infiltration for Primary Total Knee Arthroplasty
Brief Title: Liposomal Bupivacaine Versus Standard Bupivacaine Plus Dexamethasone in Quadriceps Sparing Femoral Nerve Block and Wound Infiltration for Total Knee Arthroplasty
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Eric Silverman, Director of Regional Anesthesia and Acute Pain Management, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4059
Record Dates: First submitted 2015-12-01; First posted 2015-12-09 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2016-08

CONDITIONS: Osteoarthritis; Pain, Postoperative
Keywords: primary total knee arthroplasty; liposomal bupivacaine
MeSH Terms: conditions — Osteoarthritis; Pain, Postoperative | interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposomal bupivacaine (Experimental): Liposomal bupivacaine (EXPAREL®) 133 mg in 10 mL for quadriceps sparing femoral nerve block and 133 mg in 20 mL for posterior knee compartment periarticular injection.
  Interventions: Drug: Liposomal bupivacaine
- Standard bupivacaine plus dexamethasone (Active Comparator): Bupivacaine 0.5% 10 mL plus 2 mg dexamethasone for quadriceps sparing femoral nerve block and bupivacaine 0.25% 20 mL plus 2 mg of dexamethasone for posterior knee compartment periarticular injection.
  Interventions: Drug: Bupivacaine plus dexamethasone

INTERVENTIONS:
Drug: Liposomal bupivacaine — Liposomal bupivacaine (EXPAREL®) 133 mg in 10 mL for quadriceps sparing femoral nerve block and 133 mg in 20 mL for posterior knee compartment periarticular injection.
  Arms: Liposomal bupivacaine
Drug: Bupivacaine plus dexamethasone — Bupivacaine HCl 0.5% 10 mL plus dexamethasone 2 mg for quadriceps sparing femoral nerve block and bupivacaine HCl 0.25% plus dexamethasone 2 mg for posterior knee compartment periarticular injection
  Arms: Standard bupivacaine plus dexamethasone

SUMMARY:
The purpose of this study is to compare the efficacy and duration of pain relief after total knee arthroplasty provided by a single injection of liposomal bupivacaine (EXPAREL®) versus standard bupivacaine with an adjuvant, dexamethasone when administered as a quadriceps sparing femoral nerve block and periarticular injection. It is hypothesized that liposomal bupivacaine is superior to standard bupivacaine with dexamethasone and will decrease time to discharge readiness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of American Society of Anesthesiologist (ASA) I-III physical class with a pre-operative diagnosis of primary osteoarthritis scheduled for elective primary total knee arthroplasty.
* Patients must be living independently at home prior to undergoing primary total knee arthroplasty with intention of discharge directly to home after hospitalization

Exclusion Criteria:

* Subjects will not be eligible for this trial if they have a history of allergy to a local anesthetic
* Known peripheral neuropathy
* Known connective tissue or immunological disorders
* Stroke or other known central nervous system disorders
* Renal dysfunction
* Hepatic dysfunction
* Cardiac dysfunction other than hypertension
* Pregnant subjects
* Immunosuppression
* Human immunodeficiency virus (HIV)
* Alcohol or drug abuse
* Chronic pain or opioid dependence
* Coagulopathy or those unable to comply with study requirements.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Achievement of rehabilitative goals | Time until discharge (up to 2 weeks)
  Assessment of temporal achievement of rehabilitative goals for discharge (independent ambulation to 100 feet, stair climbing, timed-up-and-go, independent toileting, ability to get dressed independently, capacity to get in and out of bed, capability to sit and rise from a chair/toilet, independence in personal care, mobilization with walker/crutches, and NRS<5 on activity).

SECONDARY OUTCOMES:
Mean postoperative pain score assessment (24, 48 and 72 hours post-operatively) | Throughout admission (up to 2 weeks)
  Assessment of mean post-operative pain using a Numeric rating scale (NRS)- both at rest and during active knee flexion to 45 degree at 24, 48 and 72 hours post-operatively.

OTHER OUTCOMES:
Cumulative pain score assessment | 24, 48 and 72 hours postoperatively
  Assessment of cumulative pain score reflected by area under the curve (AUC) for NRS scores through 12, 24, 36, 48, 60, and 72 hrs.
Mean daily Opioid consumption | 24, 48, 72 hours post-operatively, and until discharge (up to 2 weeks)
  Mean daily opioid consumption as morphine equivalents using the online calculator http://www.nyc.gov/html/doh/html/mental/MME.html
Mean length of stay in days | Through study completion (up to 2 weeks)
Time to first use of postsurgical opioid medication | Up to 24 hours postoperatively
Proportion of patients receiving no post-surgery rescue opioid medication | 0, 6, 12, 24 and 72 hours postoperatively
Discharge to home versus rehabilitation services among the comparison cohorts | Up to hospital discharge (up to 2 weeks)
Total cost comparisons between the two cohorts | Up to hospital discharge (up to 2 weeks)
  Including medications, nursing care costs, operating room costs, rehabilitation costs
Quality of recovery assessment | Postoperatively at day 0, 1, 2 and prior to discharge (up to 2 weeks)
Functional outcomes | At 6 weeks, 3 months, 6 months and 1 year postoperatively
  Functional outcomes following total knee arthroplasty at 6 weeks, 3 months, 6 months, 1 year using the Knee Society Score.
Functional outcomes | At 6 weeks, 3 months, 6 months and 1 year postoperatively
  Functional outcomes following total knee arthroplasty at 6 weeks, 3 months, 6 months, 1 year using the Lower Extremity Functional Score
Activity levels | At 6 weeks, 3 months, 6 months and 1 year postoperatively
  Activity levels following total knee arthroplasty at 6 weeks, 3 months, 6 months, and 1 year using the University of California Los Angeles scores
Objective quadriceps strength assessment | At 24 hours postoperatively
  Objective quadriceps strength assessment using a Biodex isokinetic dynamometer at 24 hours post-operatively and at the time of discharge
Patient perceived health outcomes | 6 weeks, 3 months, 6 months, and up to 1 year
  Patient perceived health outcomes at 6 weeks, 3 months, 6 months, and up to 1 year using Short Form-36 scores
Evaluate and observe any adverse reactions and complications | From time of randomization through study completion (up to 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Silverman, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

REFERENCES:
- [Background] Liu SS, Buvanendran A, Rathmell JP, Sawhney M, Bae JJ, Moric M, Perros S, Pope AJ, Poultsides L, Della Valle CJ, Shin NS, McCartney CJ, Ma Y, Shah M, Wood MJ, Manion SC, Sculco TP. Predictors for moderate to severe acute postoperative pain after total hip and knee replacement. Int Orthop. 2012 Nov;36(11):2261-7. doi: 10.1007/s00264-012-1623-5. Epub 2012 Jul 29. PMID 22842653
- [Background] Lewis C, Gunta K, Mitchell K, Bobay K. Effectiveness of multimodal pain management protocol in total knee arthroplasty patients. Orthop Nurs. 2012 May-Jun;31(3):153-9. doi: 10.1097/NOR.0b013e3182558d0b. PMID 22622607
- [Background] Barrington JW, Dalury DF, Emerson RH Jr, Hawkins RJ, Joshi GP, Stulberg BN. Improving patient outcomes through advanced pain management techniques in total hip and knee arthroplasty. Am J Orthop (Belle Mead NJ). 2013 Oct;42(10 Suppl):S1-S20. PMID 24911371
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Perlas A, Kirkham KR, Billing R, Tse C, Brull R, Gandhi R, Chan VW. The impact of analgesic modality on early ambulation following total knee arthroplasty. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):334-9. doi: 10.1097/AAP.0b013e318296b6a0. PMID 23759708
- [Background] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Background] Duellman TJ, Gaffigan C, Milbrandt JC, Allan DG. Multi-modal, pre-emptive analgesia decreases the length of hospital stay following total joint arthroplasty. Orthopedics. 2009 Mar;32(3):167. PMID 19309064
- [Background] Wang H, Boctor B, Verner J. The effect of single-injection femoral nerve block on rehabilitation and length of hospital stay after total knee replacement. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):139-44. doi: 10.1053/rapm.2002.29253. PMID 11915059
- [Background] Paul JE, Arya A, Hurlburt L, Cheng J, Thabane L, Tidy A, Murthy Y. Femoral nerve block improves analgesia outcomes after total knee arthroplasty: a meta-analysis of randomized controlled trials. Anesthesiology. 2010 Nov;113(5):1144-62. doi: 10.1097/ALN.0b013e3181f4b18. PMID 20966667
- [Background] Ng FY, Chiu KY, Yan CH, Ng KF. Continuous femoral nerve block versus patient-controlled analgesia following total knee arthroplasty. J Orthop Surg (Hong Kong). 2012 Apr;20(1):23-6. doi: 10.1177/230949901202000105. PMID 22535806
- [Background] Macfarlane AJ, Prasad GA, Chan VW, Brull R. Does regional anesthesia improve outcome after total knee arthroplasty? Clin Orthop Relat Res. 2009 Sep;467(9):2379-402. doi: 10.1007/s11999-008-0666-9. Epub 2009 Jan 7. PMID 19130163
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Kandasami M, Kinninmonth AW, Sarungi M, Baines J, Scott NB. Femoral nerve block for total knee replacement - a word of caution. Knee. 2009 Mar;16(2):98-100. doi: 10.1016/j.knee.2008.10.007. Epub 2008 Nov 28. PMID 19046884
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Background] Jaeger P, Grevstad U, Henningsen MH, Gottschau B, Mathiesen O, Dahl JB. Effect of adductor-canal-blockade on established, severe post-operative pain after total knee arthroplasty: a randomised study. Acta Anaesthesiol Scand. 2012 Sep;56(8):1013-9. doi: 10.1111/j.1399-6576.2012.02737.x. Epub 2012 Jul 26. PMID 22834681
- [Background] Ishiguro S, Yokochi A, Yoshioka K, Asano N, Deguchi A, Iwasaki Y, Sudo A, Maruyama K. Technical communication: anatomy and clinical implications of ultrasound-guided selective femoral nerve block. Anesth Analg. 2012 Dec;115(6):1467-70. doi: 10.1213/ANE.0b013e31826af956. Epub 2012 Aug 10. PMID 22886842
- [Background] Pelt CE, Anderson AW, Anderson MB, Van Dine C, Peters CL. Postoperative falls after total knee arthroplasty in patients with a femoral nerve catheter: can we reduce the incidence? J Arthroplasty. 2014 Jun;29(6):1154-7. doi: 10.1016/j.arth.2014.01.006. Epub 2014 Jan 16. PMID 24581899
- [Background] Kwofie MK, Shastri UD, Gadsden JC, Sinha SK, Abrams JH, Xu D, Salviz EA. The effects of ultrasound-guided adductor canal block versus femoral nerve block on quadriceps strength and fall risk: a blinded, randomized trial of volunteers. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):321-5. doi: 10.1097/AAP.0b013e318295df80. PMID 23788068
- [Background] Moore DC, Bridenbaugh LD, Bridenbaugh PO, Tucker GT. Bupivacaine for peripheral nerve block: A comparison with mepivacaine, lidocaine, and tetracaine. Anesthesiology. 1970 May;32(5):460-3. doi: 10.1097/00000542-197005000-00023. No abstract available. PMID 4910702
- [Background] de Leeuw MA, Dertinger JA, Hulshoff L, Hoeksema M, Perez RS, Zuurmond WW, de Lange JJ. The efficacy of levobupivacaine, ropivacaine, and bupivacaine for combined psoas compartment-sciatic nerve block in patients undergoing total hip arthroplasty. Pain Pract. 2008 Jul-Aug;8(4):241-7. doi: 10.1111/j.1533-2500.2008.00209.x. Epub 2008 May 23. PMID 18503623
- [Background] Lee AR, Yi HW, Chung IS, Ko JS, Ahn HJ, Gwak MS, Choi DH, Choi SJ. Magnesium added to bupivacaine prolongs the duration of analgesia after interscalene nerve block. Can J Anaesth. 2012 Jan;59(1):21-7. doi: 10.1007/s12630-011-9604-5. Epub 2011 Oct 20. PMID 22012543
- [Background] Naghipour B, Aghamohamadi D, Azarfarin R, Mirinazhad M, Bilehjani E, Abbasali D, Golzari SE. Dexamethasone added to bupivacaine prolongs duration of epidural analgesia. Middle East J Anaesthesiol. 2013 Feb;22(1):53-7. PMID 23833851
- [Background] Tandoc MN, Fan L, Kolesnikov S, Kruglov A, Nader ND. Adjuvant dexamethasone with bupivacaine prolongs the duration of interscalene block: a prospective randomized trial. J Anesth. 2011 Oct;25(5):704-9. doi: 10.1007/s00540-011-1180-x. Epub 2011 Jun 17. PMID 21681533
- [Background] Tripi PA, Palmer JS, Thomas S, Elder JS. Clonidine increases duration of bupivacaine caudal analgesia for ureteroneocystostomy: a double-blind prospective trial. J Urol. 2005 Sep;174(3):1081-3. doi: 10.1097/01.ju.0000169138.90628.b9. PMID 16094063
- [Background] Bailard NS, Ortiz J, Flores RA. Additives to local anesthetics for peripheral nerve blocks: Evidence, limitations, and recommendations. Am J Health Syst Pharm. 2014 Mar 1;71(5):373-85. doi: 10.2146/ajhp130336. PMID 24534592
- [Background] Williams D, Petruccelli D, Paul J, Piccirillo L, Winemaker M, de Beer J. Continuous infusion of bupivacaine following total knee arthroplasty: a randomized control trial pilot study. J Arthroplasty. 2013 Mar;28(3):479-84. doi: 10.1016/j.arth.2012.07.016. Epub 2012 Nov 2. PMID 23123039
- [Background] Beebe MJ, Allen R, Anderson MB, Swenson JD, Peters CL. Continuous femoral nerve block using 0.125% bupivacaine does not prevent early ambulation after total knee arthroplasty. Clin Orthop Relat Res. 2014 May;472(5):1394-9. doi: 10.1007/s11999-013-3164-7. PMID 23857316
- [Background] Lund J, Jenstrup MT, Jaeger P, Sorensen AM, Dahl JB. Continuous adductor-canal-blockade for adjuvant post-operative analgesia after major knee surgery: preliminary results. Acta Anaesthesiol Scand. 2011 Jan;55(1):14-9. doi: 10.1111/j.1399-6576.2010.02333.x. Epub 2010 Oct 29. PMID 21039357
- [Background] Yin C, Matchett G. Intercostal administration of liposomal bupivacaine as a prognostic nerve block prior to phenol neurolysis for intractable chest wall pain. J Pain Palliat Care Pharmacother. 2014 Mar;28(1):33-6. doi: 10.3109/15360288.2013.876485. Epub 2014 Jan 29. PMID 24476569
- [Background] Ilfeld BM, Malhotra N, Furnish TJ, Donohue MC, Madison SJ. Liposomal bupivacaine as a single-injection peripheral nerve block: a dose-response study. Anesth Analg. 2013 Nov;117(5):1248-56. doi: 10.1213/ANE.0b013e31829cc6ae. PMID 24108252
- [Background] Lonner J. Role of liposomal bupivacaine in pain management after total joint arthroplasty. J Surg Orthop Adv. 2014 Spring;23(1):37-41. doi: 10.3113/jsoa.2014.0037. PMID 24641895
- [Background] Soberon JR, Duncan SF, Sternbergh WC. Treatment of digital ischemia with liposomal bupivacaine. Case Rep Anesthesiol. 2014;2014:853243. doi: 10.1155/2014/853243. Epub 2014 Feb 5. PMID 24653844
- [Background] Bagsby DT, Ireland PH, Meneghini RM. Liposomal bupivacaine versus traditional periarticular injection for pain control after total knee arthroplasty. J Arthroplasty. 2014 Aug;29(8):1687-90. doi: 10.1016/j.arth.2014.03.034. Epub 2014 Apr 4. PMID 24793570
- [Background] Domb BG, Gupta A, Hammarstedt JE, Stake CE, Sharp K, Redmond JM. The effect of liposomal bupivacaine injection during total hip arthroplasty: a controlled cohort study. BMC Musculoskelet Disord. 2014 Sep 24;15:310. doi: 10.1186/1471-2474-15-310. PMID 25248686
- [Background] Surdam JW, Licini DJ, Baynes NT, Arce BR. The use of exparel (liposomal bupivacaine) to manage postoperative pain in unilateral total knee arthroplasty patients. J Arthroplasty. 2015 Feb;30(2):325-9. doi: 10.1016/j.arth.2014.09.004. Epub 2014 Sep 16. PMID 25282071
- [Background] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545
- [Background] McAlvin JB, Padera RF, Shankarappa SA, Reznor G, Kwon AH, Chiang HH, Yang J, Kohane DS. Multivesicular liposomal bupivacaine at the sciatic nerve. Biomaterials. 2014 May;35(15):4557-64. doi: 10.1016/j.biomaterials.2014.02.015. Epub 2014 Mar 6. PMID 24612918
- [Background] Richard BM, Newton P, Ott LR, Haan D, Brubaker AN, Cole PI, Ross PE, Rebelatto MC, Nelson KG. The Safety of EXPAREL (R) (Bupivacaine Liposome Injectable Suspension) Administered by Peripheral Nerve Block in Rabbits and Dogs. J Drug Deliv. 2012;2012:962101. doi: 10.1155/2012/962101. Epub 2012 Jan 17. PMID 22363842